CLINICAL TRIAL: NCT02035839
Title: A Pilot Multicenter Randomized Trial on the Effectiveness of Different Levels of Cooling in Comatose Survivors of Out-of-hospital Cardiac Arrest.
Brief Title: Finding the Optimal Cooling tempeRature After Out-of-HoSpiTal Cardiac Arrest
Acronym: FROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Collaborators: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FROST Trial
Record Dates: First submitted 2013-11-27; First posted 2014-01-14 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2017-05

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Target Temperature Management; Cooling comatose survivors from OHCA; Good neurological outcome at modified Rankin Score (mRS) ≤ 3
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Target Temperature Management of 34°C (Other): In hospital target temperature management to achieve core body temperature of 34°C for 24 hours.
  Interventions: Device: Target Temperature Management of 34°C
- Target Temperature Management of 32°C (Other): In hospital target temperature management to achieve core body temperature of 32°C for 24 hours.
  Interventions: Device: Target Temperature Management of 32°C
- Target Temperature Management of 33°C (Other): In hospital target temperature management to achieve core body temperature of 33°C for 24 hours.
  Interventions: Device: Target Temperature Management of 33°C

INTERVENTIONS:
Device: Target Temperature Management of 34°C — In hospital target temperature management to achieve core body temperature of 34°C for 24 hours.
  Arms: Target Temperature Management of 34°C
Device: Target Temperature Management of 32°C — In hospital target temperature management to achieve core body temperature of 32°C for 24 hours.
  Arms: Target Temperature Management of 32°C
Device: Target Temperature Management of 33°C — In hospital target temperature management to achieve core body temperature of 33°C for 24 hours.
  Arms: Target Temperature Management of 33°C

SUMMARY:
To assess the fraction of subjects surviving with good neurological outcome at 90 days for 3 different levels of hypothermia, in comatose survivors from out-of-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent (obtained from their legal representative)
* 18 years of age or older and less than 80 years old.
* Witnessed OHCA of presumed cardiac cause
* Sustained ROSC (when chest compressions have not been required for 20 consecutive minutes and signs of circulation persist)
* Initial shockable cardiac rhythm (documented by ECG or AED)
* Interval from collapse to advance life support < 20 minutes
* Interval from collapse to ROSC < 60 minutes
* Lack of meaningful response to verbal commands upon arrival to hospital after suffering non-traumatic cardiac arrest in an out-of-hospital setting
* Systolic blood pressure of >90 maintained for a least 30 minutes post-ROSC without pressors, or with a stable dose of pressors

Exclusion Criteria:

* Traumatic cardiac arrest
* Toxicological etiology
* Known or suspected pregnancy
* Do Not Attempt to Resuscitate order in force
* Unwitnessed arrest
* In-Hospital arrest
* Anatomy, previous surgery or disease state contraindicating femoral venous access
* Received neuromuscular blocking agents prior to assessing level of consciousness following ROSC
* Neurological evaluation insufficient/incomplete after ROSC but prior to randomization.
* Body core temperature < 34ºC at randomization
* Current Inferior Vena Cava (IVC) filter
* Known history of acute neurological illness or severe functional disabilities prior to arrest (e.g., seizures, traumatic brain injury, increased intracranial pressures, intra-cerebral hemorrhage, etc).
* Known hypersensitivity to hypothermia including a history of Raynaud's disease
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Terminal illness or life expectancy of less than 3 months prior to arrest
* Currently enrolled in another investigational new drug or device trial that has not completed the primary endpoint or that clinically interferes with this Trial's endpoints (For the purpose of this protocol, subjects involved in extended follow-up trials or registries for products that are currently commercially available are not considered enrolled in an investigational trial).
* Transferred from a non-participating hospital.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Fraction of subjects surviving with good neurologic outcome(modified Rankin Score (mRS) ≤ 3) at 90 days after out-of-hospital cardiac arrest. | at 90 days after out-of-hospital cardiac arrest

SECONDARY OUTCOMES:
Treatment Success: 1. proportion of subjects that can be therapeutically cooled to randomly allocated target temperature ±0.3°C (as measured by the temperature probe) | 24 hours
Treatment Success: 2. proportion of time at randomly allocated target temperature ±0.3°C during first 24 hours after initiation of induction of hypothermia | 24 hours
Treatment Success: 3. time to randomly allocated target temperature, from call to 911, sustained restoration of circulation and initiation of induction of hypothermia | 26 hours
Treatment Success: 4. rate of cooling in °C per hour | Per hour
Treatment Success: 5. rate of rewarming in °C per hour | Per hour
Outcomes: 1.Favorable neurologic status at 90 days (i.e. mRS < 3) measured as proportion | 90 days
Outcomes: 2.Time to first detected mRS ≤3 (i.e. Kaplan Meier curve) | 90 days
Outcomes: 3.Robust neurologic status at 90 days (i.e. mRS < 2) measured as proportion | 90 days
Outcomes: 4. Time to first detected mRS ≤2 (i.e. Kaplan Meier curve) | 90 days
Outcomes: 5. Survival at 90 days measured as proportion | 90 days
Outcomes: 6. Cumulative incidence of survival at 90 days (i.e. Kaplan Meier curve) | 90 days
Outcomes: 7. ICU-free survival within 90 days measured in days | 90 days
Outcomes: 8. Hospital-free survival within 90 days measured in days | 90 days
Outcomes: 9. Adverse events a. Device related b. Procedure related | 90 days
Subgroup analysis | 1 year
  A priori plan to assess heterogeneity of effect among specific subgroups of special interest as well as to assess the consistency of treatment effect among different subpopulations defined by each of multiple baseline characteristics of the patients. These will be assessed by repeating the primary analysis in the subgroups defined below, using interaction terms.
Subgroups of Special Interest Age of Patients | Duration of the trial
  18 to 65 years; or (ii) > 65 years.
Timings of initiation of hypothermia | <4 hours of restoration of spontaneous circulation; or > 4 hours
  (ii) > 65 years.
Patient Gender | Male or Female
  Subgroups to assess Consistency of Effect
Observational status of arrest | Witnessed by EMS; Witnessed by bystanders
Location of cardiac arrest | Public;Home; or Group residence (e.g. nursing home)
Bystander CPR status: | Performed; or Not performed.
AED status: | Applied by layperson;Applied by EMS provider;Not applied
Response time interval from call to initiation of CPR by EMS, among witnessed arrests: | < 10 minutes;> 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Esteban Lopez-de-Sa, M.D, Principal Investigator — Hospital Universitario La Paz. Planta
Locations (14):
- The Charité - Universitätsmedizin Berlin, Berlin, Germany
- Spain (13):
  - Hospital Universitario La Paz. Planta, Madrid, Pso. de La Castellana
  - H. Principe de Asturias, Alcalá de Henares
  - Germans Trias i Pujol University Hospital, Badalona
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañón., Madrid
  - Hospital San Carlos, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - H. University of Santiago de Compostela, Santiago de Compostela
  - Hospital Universitarion Virgen de la Macarena, Seville
  - Hospital Universitario Araba Txagorritxu, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez-de-Sa E, Juarez M, Armada E, Sanchez-Salado JC, Sanchez PL, Loma-Osorio P, Sionis A, Monedero MC, Martinez-Selles M, Martin-Benitez JC, Ariza A, Uribarri A, Garcia-Acuna JM, Villa P, Perez PJ, Storm C, Dee A, Lopez-Sendon JL. A multicentre randomized pilot trial on the effectiveness of different levels of cooling in comatose survivors of out-of-hospital cardiac arrest: the FROST-I trial. Intensive Care Med. 2018 Nov;44(11):1807-1815. doi: 10.1007/s00134-018-5256-z. Epub 2018 Oct 21. PMID 30343315